CLINICAL TRIAL: NCT04369105
Title: Influence of the Prone Position on Mechanical Power Applied to Respiratory System: Multi-centric Descriptive Study
Brief Title: Prono Position and Mechanical Power
Acronym: PROMP
Status: Completed | Type: Observational
Sponsor: Sanatorio Anchorena San Martin (Other)
Responsible Party: Principal Investigator, Matias Accoce, Head of respiratory therapists, Sanatorio Anchorena San Martin
Other Study IDs: 11/2020
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ventilation, artificial; respiratory distress syndrome, adult; prone position; monitoring, physiologic
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prone position — The patients will be put in prone position while receiving invasive mechanical ventilation and the investigators will monitor changes in mechanical power applied to the respiratory system and compare with supine position

SUMMARY:
The primary objective of the study is to compare the mechanical power applied to the respiratory system in patient with acute respiratory distress syndrome in supine positioning and after the implementation of prone positioning while mantaining the same ventilatory setting.

The secondary objetive of the study is to compare the mechanical power applied to the respiratory system in patient with acute respiratory distress syndrome in supine positioning and after the implementation of prone positioning and adjusting an individualized ventilatory setting.

DETAILED DESCRIPTION:
Data of mechanical power will be collected prospectively in three different times:

1. In supine positioning (T0).
2. After 15 minutes of having implemented prone positioning while maintaining the same ventilatory settings that in supine (T1).
3. In prone positioning after 15 min of having adjusted an individualized ventilatory setting (T2).

Besides, the investigators will take an arterial blood sample in T0 and T2 to calculate changes in oxygenation status and ventilatory ratio.

In case that esophageal manometry is available, the investigators will collect data regarding to transpulmonary and esophageal pressure in order to calculate the mechanical power applied to the lung parenchyma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged older than 18 years old under invasive mechanical ventilation with diagnostic criteria of acute respiratory distress syndrome acording to berlin definition and neccesity of prone positioning.

Exclusion Criteria:

* Need to interrump prone positioning maneuver.
* Inability to collect data for any reason.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included will be those who atend to the intensive care unit of medical centers located in Buenos Aires province, Argetina.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Mechanical power of the respiratory system measured in supine compared with prone position while maintaining the same ventilatory setting | 1) Supine position; 2) Prone position, after 15 min
  Mechanical power measured in Joules/min

SECONDARY OUTCOMES:
Mechanical power of the respiratory system measured in supine compared with prone position after adjusting the ventilatory setting | 1) Supine position; 2) Prone position, after 15 min of adjusting ventilatory setting.
  Mechanical power measured in Joules/min

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Anchorena de San Martin, San Martín, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marti J, Hall P, Hamilton P, Lamb S, McCabe C, Lall R, Darbyshire J, Young D, Hulme C. One-year resource utilisation, costs and quality of life in patients with acute respiratory distress syndrome (ARDS): secondary analysis of a randomised controlled trial. J Intensive Care. 2016 Aug 11;4:56. doi: 10.1186/s40560-016-0178-8. eCollection 2016. PMID 27525106
- [Result] Meade MO, Cook DJ, Guyatt GH, Slutsky AS, Arabi YM, Cooper DJ, Davies AR, Hand LE, Zhou Q, Thabane L, Austin P, Lapinsky S, Baxter A, Russell J, Skrobik Y, Ronco JJ, Stewart TE; Lung Open Ventilation Study Investigators. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):637-45. doi: 10.1001/jama.299.6.637. PMID 18270352
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Serpa Neto A, Deliberato RO, Johnson AEW, Bos LD, Amorim P, Pereira SM, Cazati DC, Cordioli RL, Correa TD, Pollard TJ, Schettino GPP, Timenetsky KT, Celi LA, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Mechanical power of ventilation is associated with mortality in critically ill patients: an analysis of patients in two observational cohorts. Intensive Care Med. 2018 Nov;44(11):1914-1922. doi: 10.1007/s00134-018-5375-6. Epub 2018 Oct 5. PMID 30291378
- [Result] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302